CLINICAL TRIAL: NCT05755087
Title: Phase Ib Trial of Tegavivint in Patients With Relapsed/Refractory C-MYC Overexpressing Large B-Cell Lymphoma
Brief Title: Tegavivint for Treating Patients With Relapsed or Refractory Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lapo Alinari (Other)
Responsible Party: Sponsor-Investigator, Lapo Alinari, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-21359; NCI-2023-00200 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-02-01; First posted 2023-03-06 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma Activated B-Cell Type; Recurrent Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Recurrent High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Refractory Diffuse Large B-Cell Lymphoma Activated B-Cell Type; Refractory Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Transformed Indolent B-Cell Non-Hodgkin Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Tegavivint) (Experimental): Patients receive tegavivint IV over 4 hours on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or PET and undergo blood sample collection throughout the trial. Patients may also undergo bone marrow biopsy and aspirate during screening and on the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Drug: Tegavivint; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Tegavivint — Given IV
  Other Names: BC 2059; BC-2059; BC2059; Tegatrabetan
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of bone marrow; Biopsy; Bone marrow
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of tegavivint in treating patients with large b-cell lymphomas that has come back (relapsed) or does not respond to treatment (refractory). Tegavivint may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving tegavivint may help control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of tegavivint in patients with relapsed/refractory c-Myc overexpressing large B-cell lymphoma.

II. To determine the maximum tolerated dose (MTD) or recommended phase II dose (RP2D) of tegavivint.

SECONDARY OBJECTIVES:

I. To determine the preliminary efficacy of tegavivint in patients with relapsed/refractory c-Myc overexpressing large B-cell lymphoma.

II. To determine the pharmacokinetic parameters of tegavivint.

EXPLORATORY OBJECTIVES:

I. To correlate response to tegavivint with the presence of MYC, FBW7 and SKP2 mutations.

II. To correlate response to tegavivint with TBL1 and c-Myc expression assessed by standard IHC on archived tumor biopsy.

III. To determine the effects of tegavivint on immune cell subsets viability and function.

OUTLINE: This is a dose-escalation study of tegavivint.

Patients receive tegavivint intravenously (IV) on study. Patients also undergo computed tomography (CT) and/or positron emission tomography (PET) and undergo blood sample collection throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

One of the following three conditions:

* Relapsed/refractory histologically confirmed germinal center B-cell-like (GCB) and non-GCB diffuse large B cell lymphoma (DLBCL) with the following features:

  * Increased expression of MYC (>= 40%) and BCL2 (>= 50%) by immunohistochemistry (IHC) or
  * Presence of isolated MYC translocation Or
* Relapsed/refractory histologically confirmed high-grade B-cell lymphoma (HGBCL) (double hit [DH] and triple hit [TH]) with translocations of MYC and BCL2 and/or BCL6 Or
* Histologic transformation of indolent non-Hodgkin's lymphoma (NHL) to DLBCL

  * Presence of BCL2 translocation with increased expression of MYC (≥40%) with or without MYC translocation
* Patients must have had at least two prior systemic therapies
* Patients must be ineligible for or refused autologous or allogenic hematopoietic stem cell transplantation or chimeric antigen receptor (CAR) T-cell therapy. Prior autologous stem cell transplant and/or CAR-T are allowed, if received >= 3 months prior to enrollment
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients must have radiographically measurable disease by standard positron emission tomography (PET) uptake with at least one site of measured disease by standardized uptake value (SUV)
* Absolute neutrophil count (ANC) ≥ 500/mcL
* Platelet count ≥ 25,000/mcL
* Total bilirubin =< 1.5 x the upper limit of the normal range (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 3 x institutional ULN
* Creatinine clearance >= 60 ml/min by Cockcroft-Gault (actual body weight will be used to estimate creatinine clearance)
* Patients must be willing and able to understand and give written informed consent and comply with all study related procedures
* Women of child-bearing potential (WOCBP) and men who are sexually active with WOCBP must agree to use one hormonal contraceptive (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy or tubal ligation; and one effective method of contraception, including male condom, female condom, cervical cap, diaphragm or contraceptive sponge or abstain from sex for the duration of study participation and for 4 months following completion of tegavivint administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Contraception includes:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient
* Use of oral (estrogen and progesterone), injected or implanted combined hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
* Sexually active males must use a condom during intercourse while taking drug and for 4 months after stopping study treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tegavivint or other agents used in study
* Known active central nervous system (CNS) lymphoma, history of CNS involvement allowed if in remission for >= 3 months
* Evidence of chronic active Hepatitis B, chronic active Hepatitis C infection
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy (e.g., strong CYP3A inhibitors and/or concomitant medications that are excluded) are ineligible because of the potential for pharmacokinetic interactions with tegavivint
* Known history of active TB (Bacillus Tuberculosis)
* Major surgery within 3 weeks prior to start of study treatment
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality or corrected QT interval (QTc) > 480 msec
* Uncontrolled concurrent illness including, but not limited to: ongoing or active infection (Viral, bacterial, fungal or other)
* Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and breastfeeding women are excluded from this study. The effects of tegavivint on the developing human fetus have the potential for teratogenic or abortifacient effects. There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with tegavivint
* Patients with abnormal serum chemistry values other than the specific limits detailed above, that in the opinion of the investigator is considered to be clinically significant, should be discussed with the Study PI before being enrolled in the study
* Personal history of malignancy except:

  * Cervical intraepithelial neoplasia;
  * Skin basal cell carcinoma;
  * Treated localized prostate carcinoma with prostate specific antigen (PSA) <1 ng/mL or untreated indolent prostate cancer
  * Neoplasia treated with curative intent, in remission for at least three years and considered at low risk of relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2027-03-05 (Estimated); Study Completion 2027-03-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | At the end of Cycle 1 (each cycle is 28 days)
Maximum tolerated dose (MTD) for tegavivint | At the end of Cycle 1 (each cycle is 28 days)
  Determination of the MTD of tegavivint using a 3+3 design.
Determination of the recommended phase II dose (RP2D) of tegavivint | At the end of Cycle 1 (each cycle is 28 days)

SECONDARY OUTCOMES:
Overall response rate (ORR) | After cycle 2 (each cycle is 28 days) or end of treatment
  Will be estimated by molecular subtype and across subtypes with exact 80% and 90% confidence intervals.
Complete response (CR) rate | At the end of Cycle 2 (each cycle is 28 days)
  Will be estimated by molecular subtype and across subtypes with exact 80% and 90% confidence intervals.
Duration of response (DOR) | Time from the date of first response until the first date of progression or death from any cause, assessed up to 2 years from study enrollment
  Will be summarized by the Kaplan-Meier method, and two-year estimates will be provided with 80% and 90% confidence intervals, for each subtype and for all patients.
Progression-free survival (PFS) | Time from the date of first treatment until the first date of progression or death from any cause, assessed up to 2 years from study enrollment
  Will be summarized by the Kaplan-Meier method, and two-year estimates will be provided with 80% and 90% confidence intervals, for each subtype and for all patients.
Event-free survival (EFS) | Time from the date of first treatment until the first date of progression, re-treatment of lymphoma after initial immune-therapy, or death from any cause, assessed up to 2 years from study enrollment
  Will be summarized by the Kaplan-Meier method, and two-year estimates will be provided with 80% and 90% confidence intervals, for each subtype and for all patients.
Overall survival (OS) | Time from the date of first treatment until the date of death from any cause, assessed up to 2 years from study enrollment
  Will be summarized by the Kaplan-Meier method, and two-year estimates will be provided with 80% and 90% confidence intervals, for each subtype and for all patients.

OTHER OUTCOMES:
Pharmacokinetic (PK) analysis AUC0-t | Up to 14 weeks
  The reporting of pharmacokinetic parameters will be determined based on the final parameter analysis on the available data. Parameters will be assessed using AUC0-t
Pharmacokinetic (PK) analysis AUC0-infinity | Up to 14 weeks
  The reporting of pharmacokinetic parameters will be determined based on the final parameter analysis on the available data. Parameters will be assessed using AUC0-infinity.
Pharmacokinetic (PK) analysis Tmax | Up to 14 weeks
  The reporting of pharmacokinetic parameters will be determined based on the final parameter analysis on the available data. Parameters will be assessed using Tmax
Pharmacokinetic (PK) analysis Cmax | Up to 14 weeks
  The reporting of pharmacokinetic parameters will be determined based on the final parameter analysis on the available data. Parameters will be assessed using Cmax.
Pharmacokinetic (PK) analysis t1/2 | Up to 14 weeks
  The reporting of pharmacokinetic parameters will be determined based on the final parameter analysis on the available data. Parameters will be assessed using t1/2.
Pharmacokinetic (PK) analysis clearance | Up to 14 weeks
  The reporting of pharmacokinetic parameters will be determined based on the final parameter analysis on the available data. Parameters will be assessed using clearance.
Pharmacokinetic (PK) analysis volume of distribution | Up to 14 weeks
  The reporting of pharmacokinetic parameters will be determined based on the final parameter analysis on the available data. Parameters will be assessed using volume of distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Lapo Alinari, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu